CLINICAL TRIAL: NCT04348110
Title: Evaluation of Eye Health Benefits of Blueberry Chewable Tablets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS19152
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-05

CONDITIONS: Eye

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo tablets (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo tablets
- Blueberry Chewable Tablets (Experimental)
  Interventions: Dietary Supplement: Blueberry Chewable Tablets

INTERVENTIONS:
Dietary Supplement: Placebo tablets — consume 2 tablets per day for 8 weeks
  Arms: Placebo tablets
Dietary Supplement: Blueberry Chewable Tablets — consume 2 tablets per day for 8 weeks
  Other Names: NutraView® Tablets
  Arms: Blueberry Chewable Tablets

SUMMARY:
To assess the efficacy of blueberry chewable tablets on Eye Health

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 20 years old
* Use 3C products over 6 hours per day
* Symptoms of dry eyes or tired eyes
* Tear Break-Up Time is 10 seconds less
* No history of ocular surgery (strabismus surgery, refractive surgery etc.)

Exclusion Criteria:

* Have systemic diseases affecting the front surface of the eyes.
* Long-term use of drugs or eye drops that affect the condition of the front surface of the eyes
* Long-term contact lens wear

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of Schirmer's test | 8 weeks
  Schirmer's test determines whether the eye produces enough tears to keep it moist. Units: mm (in 5minutes)
Changes of tear meniscus height | 8 weeks
  Slit lamp Ocular Surface Analyzer is utilized to measure tear meniscus height. Units: mm
Changes of non-invasive tear break-up time (NITBUT) | 8 weeks
  Ocular Surface Analyzer is utilized to measure non-invasive tear break-up time. Units: sec
Tear break-up time (TBUT) | 8 weeks
  Slit lamp ocular Surface Analyzer is utilized to measure fist tear break-up time with slit lamp. Units: sec
Changes of accommodation | 8 weeks
  Speedy-I is utilized to measure the accommodative micro fluctuation test of the ciliary muscle. Units: HFC
Ocular Surface Disease Index (OSDI) | 8 weeks
  The Ocular Surface Disease Index (OSDI) is a 12-item scale for the assessment of symptoms related to dry eye disease and their effect on vision. Units: point

SECONDARY OUTCOMES:
Changes of eye pressure | 8 weeks
  Eye pressure is measured in millimeters of mercury (mm Hg).
Changes of Intraocular pressure (IOP) | 8 weeks
  Eye pressure is measured in millimeters of mercury (mm Hg). Units: mmHg
Changes of Near point of convergence (NPC) | 8 weeks
  RAF rule were initiated in order to normalize NPC. Record as break/recovery. Units: cm
Changes of Stereo vision | 8 weeks
  The Randot Stereotest is utilized to evaluate the depth perception. Units: sec
Changes of binocular motor fusion | 8 weeks
  The test is utilized to evaluate to assess binocular motor fusion, specifically the extent to which a patient can maintain binocular single vision (BSV) in the presence of increasing vergence demands. Units: prism
Changes of Amplitude of accommodation (AA) | 8 weeks
  The amplitude of accommodation is the maximum potential increase in optical power that an eye can achieve in adjusting its focus. It refers to a certain range of object distances for which the retinal image is as sharply focused as possible. Units: diopter
Changes of Amplitude of Flipper facility | 8 weeks
  Vergence facility (VF) was measured by using a prism flipper to evaluate the ability of the fusional vergence at near with +/-2.00 flipper. Units: cpm
Changes of Fundus photography | 8 weeks
  The fundus is the back of the eye and includes the retina, optic nerve, and retinal blood vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Yie Chen, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan